CLINICAL TRIAL: NCT04066907
Title: Integrated Disease Management of Heart Failure in Primary Care; A Cluster Randomized Trial
Brief Title: Integrated Disease Management of Heart Failure in Primary Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LawsonHRI03
Record Dates: First submitted 2019-08-15; First posted 2019-08-26 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Investigator
Masking Description: A blinded research assistant will collect questionnaire data and perform NYHA assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated Disease Management (Experimental): Physicians randomized to intervention will attend a training session on the program standards and details of the IDM. Following the initial baseline interview a heart failure educator (HFE) will meet with subjects to obtain a detailed history of their HF, provide education, self-care management strategies (medication adherence, symptoms monitoring, dietary adherence, fluid restriction, exercise, weight management, smoking cessation) and review immunization status. A self-management action plan will be developed with the study physician and HFE to enable monitoring and management of HF by the participant.
  Interventions: Other: Integrated Disease Management
- Usual Care (No Intervention): Subjects will receive HF care as usually provided by their physician as advised or as needed. Study commitments for the control group include the initial interview, the expected time allotment for this initial visit is 1 hour. Telephone follow-up will occur at 3 months and 9 months to collect exacerbation data and maintain contact with participant. At 6 months and 12 months telephone follow-up will be conducted by the research assistant and the questionnaires will be completed.

INTERVENTIONS:
Other: Integrated Disease Management — Multidisciplinary intervention comprising of patient education, self management strategies and medication optimization
  Arms: Integrated Disease Management

SUMMARY:
The study population includes primary care physicians and heart failure (HF) patients attending one of over 100 family physicians in seven family health teams in Southwestern Ontario. Study purpose is to measure the effect of an integrated disease management (IDM) program for people diagnosed with HF and receiving treatment at a primary care facility. Components of IDM include HF specific patient education and self care management skills training by a heart failure educator. Study outcomes include health service use, HF symptoms, quality of life, and HF knowledge assessment compared to the usual care group.

The primary objective of this study is composite and will measure the effect of integrated disease management (IDM) on all cause hospitalizations, ED visits and mortality events. Secondary outcomes will include HF related hospitalizations, HF related ED visits, quality of life, mortality, other health service utilization, acute HF episodes, NYHA class. We hypothesize HF specific IDM implemented in primary care will be superior to usual physician-based care measured by a combined reduction in the total number of all cause hospitalizations and ED visit events.

DETAILED DESCRIPTION:
The study population will be identified through patients attending one of 100 family physicians from 10 different family health teams (FHTs) or family health organizations (FHOs) in the Southwestern Ontario.

Study Design: A parallel cluster randomized trial design has been chosen comparing the intervention arm (patients entered on the IDM) to the control arm (patients receiving usual care). A multi-level study design is proposed, level 3 the FHT/FHO, level 2 the physician and level 1 the HF patient. We have chosen to randomize at level 2, the physician and implement the intervention at both level 2 and 1, the physician and the individual. Outcomes will be measured at individual level. Stratified randomization of physicians will be performed by FHT/FHO, giving greater balance between arms and increased power and precision by reduction of between cluster variability.

Recruitment: Physicians from the FHTs/FHOs will be invited to participate and informed consent will be obtained. The physician will be randomized to either the control or intervention group and randomization will be computer generated by FHT/FHO strata. Allocation for overall study will be 1:1 as will allocation by FHT/FHO. Each participating primary care site will identify all individuals with a HF diagnosis in their care suitable for the trial and a simple random sample will be taken from this group to obtain the desired cluster size. An initial telephone call will be arranged with the patient to discuss study details, obtain informed consent, further determine eligibility, and complete questionnaires.

Data management: As a part of the objectives of this study a POSS electronic tool has been developed, all data collected about the participants will be entered by heart failure educators and stored in a central server. Access is restricted to authorized personnel only. The POSS has been designed not only as a secure storage depot but also as a tool to standardize the data collected minimizing information bias. There is extensive data checking at the time of data entry. Data definitions are incorporated to support quality data inputs.

Sample Size: With a minimum recruitment of 50 physicians recruited and 4 participants per physician, this study would be powered to detect a minimum 36% reduction in the rate of number of hospitalizations or ED visits per person year with an attrition rate of 20%. This calculation is based on 80% power to 5% significance with an ICC of 0.05.

If 100 physicians are recruited with 2 to 3 participants per physician (and a total sample size of 280) the study will have 90% power to detect a 35% reduction in the primary outcome.

Statistical Analysis: Analysis will be on an intention to treat basis. Baseline data will be used to characterize the study population, to identify any imbalances between arms. Continuous data will be displayed as mean ±standard deviation and count (percent) for categorical variables (variables to be presented will be predetermined in an analysis plan). Due to over dispersion that occurs in this type of count data the primary outcome (and health service utilization secondary outcomes) will be analyzed using a negative binomial distribution with random effects to account for clustering and for individuals experiencing multiple events. The results will be presented as rate ratios. The secondary outcomes (change in KCCQ at 6 months and other knowledge and QoL metrics) will be analyzed at individual level using logistic regression, results will be presented as odds ratios. Reliability will be assessed by using a quadrature check and in the event of failure a generalizing estimating equation (GEE) model will be fitted.

ELIGIBILITY:
Inclusion Criteria:

* New York Heart Association (NYHA) classification of stage II, III or IV
* a clinical diagnosis of HF and a supporting diagnostic echocardiogram
* HF or cardiovascular related hospitalization and/or ED visit in the 24 months prior to recruitment
* Patients with HF with a preserved ejection fraction and HF with a reduced ejection fraction (<45%) will be included.

Exclusion Criteria:

* hemodynamic instability
* awaiting cardiac surgery
* expected survival rate of <1 year due to terminal illness
* lack of English language skills
* reduced cognitive function that affects the ability to complete the questionnaires
* enrolment in other cardiac trials
* formalized HF education (e.g. Telehomecare) in the six months prior to enrolment
* scheduled for cardiac rehabilitation
* severely impaired renal function requiring dialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2024-08-05 (Estimated); Study Completion 2024-08-05 (Estimated)

PRIMARY OUTCOMES:
Composite of all cause mortality, hospital admissions and emergency department visits | 1 year
  The primary outcome will be a composite of the total number of all-cause mortality, hospital admissions, and ED visits events. This measure will be the rate of events per person year at risk. The ED visits will be visits that do not lead to hospitalization.

SECONDARY OUTCOMES:
Quality of Life using KCCQ | 6 months and 1 year
  Quality of life measure using the Kansas City Cardiomyopathy Questionnaire (KCCQ). The KCCQ is a self-administered questionnaire that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. An improvement in total score will indicate an improvement in health status and quality of life. The range is score is from 0-100
Mortality | 1 year (rate number of events per person year of follow-up)
  All cause mortality rate
Health Status using EQ-5D | 6 months and 1 year
  Measure health status of health for clinical and economic appraisal using the EQ-5D. The EQ-5D is a self-administered questionnaire and is comprised of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. An decrease in total score will indicate an improvement in health status. The range of the scale is from 5-25.
Health Status using SF-12 | 6 months and 1 year
  Measure overall health status using the SF-12. The SF-12 is a self-administered questionnaire that measures physical and mental health composite scores with twelve questions that range from 0-100. An improvement in score will indicate an improvement in health status.
Health Service Use - Hospitalization | 1 year (rate number of events per person year of follow-up)
  Number of heart failure related hospitalizations during study. Number of all-cause hospitalizations during study.
Health Service Use - Emergency Department visit | 1 year (rate number of events per person year of follow-up)
  Number of heart failure related emergency department visits. Number of all-cause emergency department visits during study.
Atlanta Heart Failure Knowledge Questionnaire | 1 year
  The Atlanta Heart Failure Knowledge Questionnaire (AHFKQ) consists of 30 questions and was developed to ascertain knowledge about HF, treatment, and self-care.
The Mediterranean Diet Questionnaire | 1 year
  The Mediterranean Diet is a 14-item questionnaire to assess adhesion to a Mediterranean diet, proven to be beneficial to people with heart failure
NYHA | 1 year
  NYHA: The NYHA is a classification system for the extent of HF. It classifies patients in one of four categories based on limitations during physical activity due to symptoms of HF
Health Service Use -unscheduled physician visits | 1 year (rate number of events per person year of follow-up)
  Number of heart failure related unscheduled physician visits
Health Service Use -urgent care facility visits | 1 year (rate number of events per person year of follow-up)
  Number of heart failure related urgent care facility visits
Acute Heart Failure Episodes | 1 year (rate number of events per person year of follow-up)
  An acute HF episode will be recorded if the participant experiences any of the following:
  i. Worsening signs or symptoms of HF leading to an unscheduled physician visit and/or urgent care facility.
  ii. Worsening signs or symptoms of HF leading to a visit to an ED. iii. Worsening signs or symptoms of HF leading to hospitalization. iv. Worsening signs or symptoms of HF leading to an activation of action plan

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Licskai, Principal Investigator — Lawson
Locations (1):
- London Health Science Center, Victoria Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hussey AJ, McKelvie RS, Ferrone M, To T, Fisk M, Singh D, Faulds C, Licskai C. Primary care-based integrated disease management for heart failure: a study protocol for a cluster randomised controlled trial. BMJ Open. 2022 May 12;12(5):e058608. doi: 10.1136/bmjopen-2021-058608. PMID 35551078